CLINICAL TRIAL: NCT00003004
Title: An Open-Label, Non-Randomized Phase I Study of the Protein Kinase C Inhibitor Flavopiridol Administered in Combination With Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Refractory or Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 96-077; CDR0000065571 (Registry Identifier: PDQ (Physician Data Query)); NCI-T96-0091
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — alvocidib; Cisplatin; Paclitaxel

INTERVENTIONS:
Drug: alvocidib
Drug: cisplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy with paclitaxel and cisplatin plus flavopiridol in treating patients who have refractory or recurrent solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of flavopiridol when administered in combination with paclitaxel and cisplatin in patients with refractory adult solid tumors. II. Investigate the clinical pharmacokinetics of intravenous flavopiridol when administered in combination with paclitaxel in these patients. III. Obtain preliminary data on the therapeutic activity of flavopiridol when administered in combination with paclitaxel in these patients. IV. Evaluate surrogate markers of activity such as inhibition of PKC or CDK1 in these patients.

OUTLINE: This is an open label, dose escalation study. Patients receive paclitaxel IV over 3 hours on day 1. On day 2, patients receive cisplatin IV over 20 minutes followed by a 24 hour infusion of flavopiridol. Courses are repeated every 21 days in the absence of disease progression or unacceptable toxicity. Sequential dose escalation of flavopiridol is followed by sequential dose escalation of cisplatin. Dose escalation in cohorts of 3-6 patients each continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity. Patients are followed every 6 weeks.

PROJECTED ACCRUAL: Approximately 46-73 patients will be accrued for this study within 6 more months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven solid tumors that are refractory or recurrent -No CNS primary or metastatic disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance Status: Karnofsky at least 60% Hematopoietic: WBC at least 3,500/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL AST and ALT no greater than 2.5 times upper limit of normal Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: At least 6 months since prior cardiac arrhythmias, myocardial infarction, or congestive heart failure Other: Not pregnant or nursing Effective contraceptive method must be used for 2 months after study completion Not HIV positive No uncontrolled or serious infection No pre-existing grade 3 or greater neurotoxicity Must be mentally capable of understanding the explanation of the study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior immunotherapy Chemotherapy: At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy Surgery: Not specified Other: No presence of toxic effects from prior therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 1997-07; Primary Completion 2001-10 (Actual); Study Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States